## Autologous Hematopoietic System Cell Transplant for Patients with Systemic Sclerosis and Cardiac Dysfunction NCT03593902 10/09/2019

## Statistical Methods

Continuous variables (as age, FVC, TLC, DLCO, PASP, and mPAP) to be summarized as means and standard deviations and their differences between groups to be assessed via the Wilcoxon rank-sum test. Categorical variables (as sex and relapse) to be summarized as counts and proportions, and differences in categorical variables between groups to be assessed via Fisher's exact test.